CLINICAL TRIAL: NCT04743635
Title: CONtrolled Focal Fibrous Band Release Method Study
Acronym: CONFFIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revelle Aesthetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-10472
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-06

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Intervention Model Description: All participants were treated with the Avéli device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Targeted Verifiable Subcision (TVS) with the Avéli device, mITT (Experimental): Modified intent to treat population (n=68). The modified intent to treat population was used to evaluate effectiveness.
  The single procedure was conducted using the Avéli device for TVS. Cellulite can be treated on the thighs and buttocks
  Interventions: Device: Avéli device
- Targeted Verifiable Subcision (TVS) with the Avéli device, Roll-in (Experimental): The roll-in population (n=6) was excluded from the effectiveness analyses. For Investigators that have not previously performed an Avéli procedure, two (2) participants were classified as roll-in participants. The single procedure was conducted using the Avéli device for TVS. Cellulite can be treated on the thighs and buttocks
  Interventions: Device: Avéli device

INTERVENTIONS:
Device: Avéli device — Minimally invasive single procedure with the Avéli device for reduction in the appearance of cellulite in the thighs and buttocks.

SUMMARY:
Study to evaluate the safety and effectiveness of the Avéli medical device to reduce the appearance of cellulite.

DETAILED DESCRIPTION:
Multi-center, single-arm clinical study to evaluate the safety and effectiveness of the Avéli device in reducing the appearance of cellulite.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe cellulite

Exclusion Criteria:

* Body Mass Index ≥30.0

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. G. William Stevens, MD, Principal Investigator — Marina Plastic Surgery
Locations (9):
- United States (7):
  - Clinical Site #3, Los Angeles, California
  - Clinical Site #5, San Diego, California
  - Clinical Site #4, San Francisco, California
  - Clinical Site #2, Coral Gables, Florida
  - Clinical Site #6, Shreveport, Louisiana
  - Clinical Site #8, Chestnut Hill, Massachusetts
  - Clinical Site #1, Minneapolis, Minnesota
- Australia (2):
  - Clinical Site #7, Southport, Queensland
  - Clinical Site #9, Toowoomba, Queensland

IPD SHARING:
Plan to Share IPD: Yes
Plan to share Executive Summary of Protocol. No formal, separate SAP for this study.
Supporting Information: Study Protocol
Time Frame: Will post Protocol Executive Summary on June 14, 2022. It will be available indefinitely.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 was total enrollment:
  * 68 participants allocated to Targeted Verifiable Subcision (TVS) with the Avéli device, mITT
  * 6 participants allocated to Targeted Verifiable Subcision (TVS) with the Avéli device, Roll-Ins. 6 training participants for 3 new Investigators.
Groups:
- Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT: N=68, included in the effectiveness analyses Allocation: non-randomized Intervention Model: Single Group Assignment
- Targeted Verifiable Subcision (TVS) With the Avéli Device, Roll-in: N=6, excluded from the effectiveness analyses. The first two participants treated by three Investigators who never used the Avéli device were classified as roll-ins.
  Allocation: non-randomized Intervention model: Single group assignment
Period: Overall Study
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT | Targeted Verifiable Subcision (TVS) With the Avéli Device, Roll-in
Started | 68 | 6
Completed | 66 | 6
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Targeted Verifiable Subcision (TVS) With the Avéli Device: Modified intent to treat population (mITT), n=68. Cellulite can be treated across thighs and buttocks. Minimally invasive procedure: Procedure for reducing cellulite.
- Targeted Verifiable Subcision (TVS) With the Avéli Device, Roll-in: Roll-in participants, n=6. Cellulite can be treated across thighs and buttocks. Minimally invasive procedure: Procedure for reducing cellulite.
- Total: Total of all reporting groups
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device | Targeted Verifiable Subcision (TVS) With the Avéli Device, Roll-in | Total
Number analyzed (Participants) | 68 | 6 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (7.4) | 40.8 (8.1) | 41.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 6 | 74
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 2 | 21
  Not Hispanic or Latino | 49 | 4 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 0 | 6
  White | 54 | 6 | 60
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 52 | 6 | 58
  Australia | 16 | 0 | 16
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Used by site to evaluate the participant's skin type using the following scale:
  Type 1: light, pale white Type 2: white, fair Type 3: medium white to olive Type 4: olive, moderate brown Type 5: brown, dark brown Type 6: black, very dark, brown to black
  Participants
    I | 1 | 2 | 3
    II | 19 | 1 | 20
    III | 24 | 2 | 26
    IV | 15 | 1 | 16
    V | 6 | 0 | 6
    VI | 3 | 0 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.9 (2.6) | 23.1 (3.6) | 24.8 (2.7)
Laxity [Count of Participants; unit: Participants]
  None | 1 | 0 | 1
  Mild | 37 | 3 | 40
  Moderate | 30 | 3 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Mean Change From Baseline to 3 Months in Cellulite Severity Scale (CSS) Score for Participants
Description: The CSS includes a 6-point (range of 0-5) and will be determined by 3 independent, blinded physician assessors of images obtained before and 3-months after treatment.
  CSS Scale TOTAL CSS SCORE: = (PART A + PART B) - 1
  PART A- Number of evident depressions 0 None
  1. Mild (≤4 depressions)
  2. Moderate (5 to 9 depressions)
  3. Severe (≥ 10 depressions) PART B - Average depth of depressions
  0 None
  1. Mild (1-2 mm)
  2. Moderate (3-4 mm)
  3. Severe (≥5 mm)
Time Frame: 3 months
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT: Allocation: N/A, Intervention Model: Single Group Assignment
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT
Number analyzed (Participants) | 68
score on a scale | 1.5 (0.9)
Statistical Analysis 1: Comparison: Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT; The endpoint tested the mean of the changes for each treated participant, not a 1-point change between mean score of the group at baseline versus 3 months. Success is achieved when the mean change across all treated participants is at least one point; Test type: Other — Performance goal. Hypothesis: Ho: D < 1 Ha: D ≥ 1, where D = reduction in the CSS score from baseline to 3 months, and 1 is the performance goal. If the lower bound of the two-sided 95% confidence interval is greater than or equal to 1 then we will reject the null hypothesis and conclude the device performs effectively; p = .0001, t-test, 2 sided; The 2-sided 95% confidence interval for the mean reduction in CSS was calculated along with the corresponding p-value (Student's t-test); Mean Difference (Final Values) = 1.5, 95% CI 2-sided [1.28 to 1.71], Standard Deviation .9

2. Secondary Outcome: Percentage of Participants With Improvement as Assessed Using Global Aesthetic Improvement Scale (GAIS) at 3 Months
Description: The GAIS score was determined by blinded, independent evaluators. The GAIS scale counted if at least two of the three evaluators selected it, otherwise the median between the three was counted. A participant is considered improved if the GAIS assessment is improved (1), much improved (2) or very much improved (3). The hierarchal endpoint is met if the lower bound of the 2-sided 95% confidence interval is greater than or equal to 0.6.
  Scale: -3:very much worse, the treated area appearance is worse than before procedure, -2: much worse, the treated area appearance is significantly worse than before procedure, -1: worsened, the treated area appearance is slightly worse than before procedure, 0:no change, the treated area appearance is the same, +1: improved, noticeable improvement in appearance of the treated areas, but subtle, +2: much improved, significant improvement in appearance in the treated areas, +3: very much improved, optimal cosmetic result in the treated areas.
Time Frame: 3 months
Population: mITT
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT
Number analyzed (Participants) | 68
Percentage of participants | 95.6 [87.6 to 99.1]
Statistical Analysis 1: Comparison: Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT; The GAIS scale counted if at least two of the three evaluators selected it, otherwise the median between the three was counted (e.g., if "improved", "worse" and "much worse", "worse" was counted). A participant is considered improved if the GAIS assessment is improved (1), much improved (2) or very much improved (3); Test type: Other — Performance goal. The hierarchal endpoint is met if the lower bound of the 2-sided 95% confidence interval is greater than or equal to 0.6; p = .0001, t-test, 2 sided; Percentage improved = 95.6, 95% CI 2-sided [87.6 to 99.1]

3. Secondary Outcome: Percentage of Participants With Improvement as Assessed Using Global Aesthetic Improvement Scale (GAIS) at 12 Months
Description: The GAIS score was determined by blinded, independent evaluators. The GAIS scale counted if at least two of the three evaluators selected it, otherwise the median between the three was counted. A participant is considered improved if the GAIS assessment is improved (1), much improved (2) or very much improved (3).
  Scale: -3: very much worse, the treated area appearance is worse than before procedure, -2: much worse, the treated area appearance is significantly worse than before procedure, -1: worsened, the treated area appearance is slightly worse than before procedure, 0:no change, the treated area appearance is the same, +1: improved, noticeable improvement in appearance of the treated areas, but subtle, +2: much improved, significant improvement in appearance in the treated areas, +3: very much improved, optimal cosmetic result in the treated areas.
Time Frame: 12 Months
Population: mITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT
Number analyzed (Participants) | 65
percentage of participants | 93.85 [84.99 to 98.30]

4. Secondary Outcome: The Mean Change From Baseline to 12 Months in Cellulite Severity Scale (CSS) Score for Participants
Description: as for outcome 1
Time Frame: 12 months
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT
Number analyzed (Participants) | 65
score on a scale | 1.48 (0.87)

5. Secondary Outcome: The Percentage of Patients Satisfied With Their Results at 3 Months
Description: Participants were asked to rate their satisfaction with their results (from very satisfied to very dissatisfied) in an online questionnaire at 3 months. The outcome measure reports the percentage of participants satisfied with their results at 3 months. The Site was blinded to the questionnaire data. The sponsor was only unblinded after the data analyses.
  The lower bound of the 2-sided 95% confidence interval had to be greater than or equal to 0.6.
Time Frame: 3 month
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT
Number analyzed (Participants) | 68
percentage of participants | 72.1 [59.9 to 82.3]
Statistical Analysis 1: Comparison: Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT; Test type: Other — Performance goal. In order to meet the endpoint, the lower bound of the 2-sided 95% confidence interval had to be greater than or equal to 0.6; p = .0264, t-test, 2 sided; Percentage improved = 72.1, 95% CI 2-sided [59.9 to 82.3]

6. Secondary Outcome: The Number of Patients Satisfied With Their Results at 12 Months
Description: Participants were asked to rate their satisfaction with their results (from very satisfied to very dissatisfied) in an online questionnaire at 12 months. The outcome measure reports the number of participants satisfied with their results at 12 months. The Site was blinded to the questionnaire data. The sponsor was only unblinded after the data analyses.
Time Frame: 12 Months
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT
Number analyzed (Participants) | 65
Participants | 45

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events (AEs) were defined as any undesirable medical occurrence providing the most comprehensive, real-world safety profile. This definition does not depend on a causal relationship with the device. At each visit, the investigator determined whether any AEs occurred. The Medical Monitor reviewed all adverse events and assigned the MedDRA lower-level term (LLT) codes. The Common Terminology Criteria for Adverse Events (CTCAE) scale grades 1-5 was used in CONFFIRM to describe AE severity.
Groups:
- Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT: Modified intent to treat population (mITT), n=68. Cellulite can be treated across thighs and buttocks. Minimally invasive procedure: Procedure for reducing cellulite.
Arm/Group | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT | Targeted Verifiable Subcision (TVS) With the Avéli Device, Roll-in
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/6
Other Adverse Events (participants affected / at risk) | 68/68 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted Verifiable Subcision (TVS) With the Avéli Device, mITT (N=68) | Targeted Verifiable Subcision (TVS) With the Avéli Device, Roll-in (N=6)
Ecchymosis (Skin and subcutaneous tissue disorders) | 59 (59) | 6 (6)
Tenderness (General disorders) | 35 (35) | 3 (3)
Pain (General disorders) | 26 (26) | 2 (2)
Induration (General disorders) | 25 (25) | 2 (2)
Incision site bleeding (General disorders) | 11 (11) | 0 (0)
Numbness (Nervous system disorders) | 12 (12) | 0 (0)
Edema (General disorders) | 8 (8) | 1 (1)
Fluid Discharge (General disorders) | 6 (6) | 0 (0)
Hemosiderin stain (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Swelling (General disorders) | 4 (4) | 0 (0)
Burning sensation (General disorders) | 3 (3) | 0 (0)
Tingling (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) — Hyperpigementation of skin
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT04743635/Prot_SAP_000.pdf